CLINICAL TRIAL: NCT00263757
Title: A Randomized Trial of Positive Airway Pressure Therapy In Atrial Fibrillation Recurrence In Sleep Apnea
Brief Title: Atrial Fibrillation Recurrence in Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH); ResMed Foundation (Other)
Responsible Party: Sean M. Caples, D.O, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1254-05; 1RC1HL099534 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Sleep Apnea; Atrial Fibrillation
MeSH Terms: conditions — Sleep Apnea Syndromes; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic Positive Airway Pressure (Experimental): Subjects randomized to this arm received nightly Adaptive Servo-Ventilation during sleep for 12 months.
  Interventions: Device: Adaptive Servo-Ventilation
- Usual Care (Other): Subjects randomized to this arm received medical management for 12 months as prescribed by their cardiologist.
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Adaptive Servo-Ventilation — Adaptive Servo-Ventilation provides positive expiratory airway pressure and inspiratory pressure support, which is servocontrolled based on the detection of central sleep apnea.
  Arms: Therapeutic Positive Airway Pressure
Other: Usual Care — Subjects randomized to this arm received medical management as prescribed by their cardiologist.
  Arms: Usual Care

SUMMARY:
This randomized, controlled trial is designed to test whether treatment of sleep disordered breathing (SDB) with positive airway pressure (PAP) therapy alters the natural history of atrial fibrillation (AF). Patients with recent AF who are now in sinus rhythm, and found to have SDB (obstructive and/or central sleep apnea) by formal sleep study but without complaints of daytime sleepiness, are randomized to PAP therapy to eradicate SDB or to usual care (medical management as prescribed by the patient's cardiologist).

DETAILED DESCRIPTION:
Sleep apnea is a common disorder which is increasingly implicated in the pathogenesis of cardiovascular disease. Observational data suggest that sleep apnea may play a role in the development of atrial fibrillation (AF), and may even predispose to recurrence of AF following electrical cardioversion (DCCV). Because of biases and confounders inherent to observational studies, we propose a randomized clinical trial to assess the effects of treatment of sleep apnea in subjects with AF treated with DCCV. Following polysomnography, subjects with sleep apnea will be randomized to positive airway pressure (PAP) or usual medical care and followed for up to one year to compare a primary outcome of AF recurrence rate.

ELIGIBILITY:
Inclusion criteria:

1. Age >18 yrs
2. Successful electrical or chemical cardioversion within previous 2 weeks
3. Greater than 2 episodes symptomatic AF in previous 6 months

Exclusion criteria:

1. Currently on PAP therapy
2. Moderate to severe pulmonary disease
3. Neurologic impairment (h/o cerebrovascular accident (CVA), transient ischemic attack (TIA), neuromuscular disease, diaphragmatic paralysis)
4. Severe cardiac disease (LVEF<40%, greater than mild to moderate valvular disease)
5. Post cardiac surgery AF
6. Congenital heart disease
7. Renal disease (Scr > 2.5)
8. Excessive ethanol (EtOH) use (>2 drinks/day)
9. Anatomically fixed nasal obstruction (severe septal deviation, uncontrolled rhinitis)
10. History of motor vehicle or occupational accident related to sleepiness.
11. Epworth Sleepiness Scale score >18 (out of maximum score of 24).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean M. Caples, D.O., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Caples SM, Mansukhani MP, Friedman PA, Somers VK. The impact of continuous positive airway pressure treatment on the recurrence of atrial fibrillation post cardioversion: A randomized controlled trial. Int J Cardiol. 2019 Mar 1;278:133-136. doi: 10.1016/j.ijcard.2018.11.100. Epub 2018 Nov 20. PMID 30522886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care
Started | 12 | 13
Completed | 4 | 5
Not Completed | 8 | 8
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Screen failure | 0 | 1
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had Atrial Fibrillation Recurrence at 1 Year
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care
Number analyzed (Participants) | 12 | 13
participants | 3 | 3

2. Secondary Outcome: Mean Score on Epworth Sleepiness Scale (ESS) at Baseline and 12 Month Visit
Description: The ESS is a measure of general level of sleepiness. The ESS asks subjects to rate their usual chances of dozing off or falling asleep in 8 different situations or activities that most people engage in as part of their daily live, although not necessarily every day. The questionnaire has 8 questions, with responses ranging from 0 (would never dose) to 3 (high chance of dozing). Therefore the total score could range from 0 (no sleepiness) to 24 (high chance of dozing).
Time Frame: baseline, 12 months
Population: Usual Care Arm: At the baseline visit 13 participants completed the ESS, and at the 12 month visit 6 participants completed the ESS, due to withdrawals.
  Therapeutic Positive Airway Pressure Arm: At the baseline visit 12 participants completed the ESS, and at the 12 month visit 5 participants completed the ESS, due to withdrawals.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline Visit, n=12, 13 | 4.75 (2.14) | 7.31 (3.33)
  12 Month Visit, n=5, 6 | 5.80 (2.59) | 5.67 (2.34)

3. Secondary Outcome: Mean Score on Functional Outcomes of Sleep Questionnaire (FOSQ)
Description: The FOSQ is a disease-specific quality of life questionnaire to determine functional status in adults. The measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living. There are 30 items on the questionnaire consisting of 5 factor subscales. The subject rates the difficulty of performing a given activity on a 4-point scale (no difficulty to extreme difficulty). A higher score indicates greater difficulty or impact of sleepiness on daily living. FOSQ total score ranges from 0 (no difficulty) to 120 (extreme difficulty).
Time Frame: baseline, 12 months
Population: Usual Care Arm: At the baseline visit 13 participants completed the FOSQ, and at the 12 month visit 4 participants completed the FOSQ, some due to withdrawals.
  Therapeutic Positive Airway Pressure Arm: At the baseline visit 12 participants completed the FOSQ, and at the 12 month visit 4 participants completed the FOSQ, due to withdrawals.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline visit, n=12, 13 | 19.08 (0.67) | 17.62 (1.56)
  12 months visit, n=4, 4 | 18.25 (1.50) | 17.50 (1.91)

ADVERSE EVENTS:
Arm/Group | Therapeutic Positive Airway Pressure | Usual Care
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/13
Other Adverse Events (participants affected / at risk) | 1/12 | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Positive Airway Pressure (N=12) | Usual Care (N=13)
Interim hospitalization (General disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Positive Airway Pressure (N=12) | Usual Care (N=13)
Worsening breathlessness during the day (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Worsening breathlessness/gasping awaken from sleep (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chest pain at night/awakens from sleep (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary barrier to enrollment was the high rate of subjects who were previously diagnosed with sleep apnea and were already prescribed treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No